CLINICAL TRIAL: NCT03598543
Title: Klebsiella Pneumoniae Infection in China: Epidemiology, Molecular Characteristics, Treatment, and Outcome
Brief Title: Epidemiology of Klebsiella Pneumoniae in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Jian-cang Zhou M.D., Prof., Sir Run Run Shaw Hospital
Other Study IDs: SRRSH-China-KP
Record Dates: First submitted 2018-07-15; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Klebsiella Pneumoniae Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Carbapenem-Sensitive K. pneumoniae: Any patients with clinical confirmed Carbapenem-Sensitive Klebsiella pneumoniae infection.
  Interventions: Other: no intervention
- Carbapenem-Resistant K. pneumoniae: Patients with clinical confirmed Carbapenem-Resistant Klebsiella pneumoniae infection.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention, this is an obervational study.

SUMMARY:
Klebsiella pneumoniae is one of the most common pathogens causing both community-onset and nosocomial infection. More worse, the emergency of Carbapenem-Resistant Klebsiella pneumoniae (CRKP) had cause the clinical therapy be very difficult. However, there is not much empirical data as to the prevalence, risk factors, characteristics,outcomes and the rationality of the current therapy for the Klebsiella pneumoniae infection in China.Thus, the study was aimed to investigate the epidemiology and risk factors, characteristics, outcomes and the rationality of the current therapy for the Klebsiella pneumoniae infection in China.

DETAILED DESCRIPTION:
All the patients with culture positive of Klebsiella pneumoniae were screened and reported to the the clinical doctors and confirmed by them. And the clinical characteristics of the patiens, such as baseline data, outcomes etc, were recorded. Finially, to find the prevalence, risk factors, characteristics, outcome and the rationality of the current therapy for the Klebsiella pneumoniae infection in China.

ELIGIBILITY:
Inclusion Criteria:

- new confirmed community-onset or noscomial infection of Klebsiella pneumoniae infection

Exclusion Criteria:

* Age<18, or >85 years old; Mixed infection of Klebsiella pneumoniae and other microbes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patients with the age between 18 and 85 years old and with either community or hospital Klebsiella pneumoniae infection.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
CRKP infection | 6 months
  Culture postitive results confirmed the infection of CRKP

CONTACTS AND LOCATIONS:
Overall Officials: Yun-song Yu, MD, Principal Investigator — Zhejiang University
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided